CLINICAL TRIAL: NCT04513951
Title: Phase II Study of AVELUMAB and CETUXIMAB and Modified FOLFOXIRI as Initial Therapy for RAS Wild-type Unresectable Metastatic Colorectal Cancer Patients
Brief Title: AVELUMAB and CETUXIMAB and mFOLFOXIRI as Initial Therapy for Unresectable Metastatic Colorectal Cancer Patients
Acronym: AVETRIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001501-24
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: modified FOLFOXIRI; Cetuximab; Avelumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Irinotecan; Oxaliplatin; Cetuximab; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mFOLFOXIRI + Cetuximab + Avelumab (Experimental): * Avelumab, 800 mg intravenous [IV] dose over 60 minutes, day 1, followed by
  * Cetuximab, 500 mg/m2 IV dose over 2 hours at cycle 1 (if well tolerated, it is administered over 90 minutes at cycle 2 and over 60 minutes by cycle 3), day 1, followed by
  * Irinotecan 150 mg/ m2 IV dose over 60 minutes day 1, followed by
  * Oxaliplatin 85 mg/m2 IV dose over 2 hours, day 1 in two-way with
  * L-Leucovorin 200 mg/ m2 IV dose over 2 hours, day 1 followed by
  * 5-fluoruracil 2400 mg/m2 IV dose 48 h-continuous infusion, starting on day 1; to be repeated every 14 days for a maximum of 12 cycles. If no progression occurs during the induction treatment, patients will receive maintenance with 5-FU/LV plus cetuximab and avelumab at the same dose used at the last cycle of the induction treatment. 5-FU/LV plus cetuximab and avelumab will be repeated biweekly until disease progression, unacceptable toxicity, patient's refusal or consent withdrawal.
  Interventions: Drug: 5Fluorouracil; Drug: L-leucovorin; Drug: Irinotecan; Drug: Oxaliplatin; Drug: Cetuximab; Drug: Avelumab

INTERVENTIONS:
Drug: 5Fluorouracil — phase II
Drug: L-leucovorin — phase II
Drug: Irinotecan — phase II
Drug: Oxaliplatin — phase II
Drug: Cetuximab — phase II
Drug: Avelumab — phase II

SUMMARY:
The aim of this study is to evaluate the efficacy of mFOLFOXIRI plus cetuximab and avelumab as first line treatment of patients with initially unresectable and previously untreated RAS wild-type metastatic colorectal cancer (mCRC), in terms of Progression-free Survival.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicentric phase II single-arm trial in which patients with initially unresectable and previously untreated RAS wild-type mCRC will receive induction treatment with mFOLFOXIRI plus cetuximab and avelumab up to 12 cycles followed by maintenance with 5-FU/LV plus cetuximab plus avelumab until disease progression, unacceptable toxicity or patient's refusal. The second- and subsequent lines of treatment will be at investigators' choice.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of colorectal adenocarcinoma;
* Initially unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease;
* At least one measurable lesion according to RECIST 1.1.;
* Availability of a tumour tissue sample (primary tumour and/or metastatic sites);
* Male or female of 18-75 years of age;
* ECOG PS ≤2 for patients aged ≤70 years; ECOG PS 0 for patients aged 71 to 75 years;
* Life expectancy of at least 12 weeks;
* Previous adjuvant chemotherapy allowed only if with fluoropyrimidine monotherapy and more than 6 months elapsed between the end of adjuvant and first relapse;
* RAS (codons 12, 13, 59, 61, 117 and 146 of KRAS and NRAS genes) wild-type status of primary colorectal cancer or related metastasis (local or central laboratory assessment);
* Adequate haematological function: neutrophils >1.5 x 109/L, platelets >100 x 109/L, haemoglobin >9 g/dl;
* Adequate liver and renal function: total bilirubin 1.5 time the upper-normal limits (UNL) of the normal values and AST (SGOT) and/or ALT (SGPT) <2.5 x UNL (or <5 x UNL in case of liver metastases) alkaline phosphatase <2.5 x UNL (or <5 x UNL in case of liver metastases); creatinine clearance ≥50 mL/min or serum creatinine 1.5 x UNL;
* INR or aPTT ≤1.5 × ULN. Patients who are on therapeutic doses of anti-coagulants are eligible if they are on a stable dose of anti-coagulant for 28 days with stable INR and PTT values;
* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 continuous months, are surgically sterile, or are sexually inactive;
* Subjects and their partners must be willing to avoid pregnancy during the trial and until 6 months after the last trial treatment. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception as approved by the investigator (barriere contraceptive measure or oral contraception);
* Will and ability to comply with the protocol;
* Written informed consent to study procedures and to molecular analyses.

Exclusion Criteria:

* Radiotherapy to any site within 4 weeks before the study;
* Previous adjuvant oxaliplatin-containing chemotherapy;
* Previous treatment with cetuximab;
* Prior treatment with CD137 agonists, anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents;
* Treatment with any investigational drug within 30 days prior to enrollment or 2 investigational agent half-lives (whichever is longer);
* Major surgery for any reason, except diagnostic biopsy, within 4 weeks of the trial treatment and/or if the subject has not fully recovered from the surgery within 4 weeks of the trial treatment, or anticipation of the need for major surgical procedure during the course of the study;
* Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of the trial treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement dose, equivalent to < 10 mg prednisone daily).

Notes:

1. Subjects receiving bisphosphonate or denosumab are eligible provided treatment was initiated at least 14 days before first dose of trial treatment;
2. Previous or ongoing administration of systemic steroids for the management of an acute allergic phenomenon is acceptable as long as it is anticipated that the administration of steroids will be completed in 14 days, or that the daily dose after 14 days will be ≤ 10 mg per day of equivalent prednisone.

   * All subjects with brain metastases, except those meeting the following criteria:

a. Brain metastases have been treated locally, have not been progressing at least 2 months after completion of therapy, and no steroid maintenance therapy is required, and b. No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable).

* Symptomatic peripheral neuropathy > 2 grade NCI-CTCAE v5.0;
* Other co-existing malignancies or previous malignant disease (other than colorectal cancer) within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or carcinoma in situ (bladder, cervical, breast);
* Prior organ transplantation, including allogeneic stem cell transplantation;
* Significant acute or chronic infections, including, among others:

  1. Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome;
  2. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test prior to registration) or hepatitis C. Notes: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
  3. Active tuberculosis (history of exposure or history of positive TB test; plus presence of clinical symptoms, physical or radiographic findings).
* Active autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, that might deteriorate when receiving an immunostimulatory agent:

  1. Subjects with diabetes type I, vitiligo, psoriasis, hypo- and hyperthyroid disease not requiring immunosuppressive treatment are eligible;
  2. History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study;
  3. History of controlled type I diabetes mellitus on a stable insulin regimen may be eligible for this study;
  4. Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at dose ≤ 10 mg or 10 mg equivalent prednisone per day;
  5. Administration of steroids through a route known to result in minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable.
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan. Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted;
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to moAbs (NCI CTCAE v5.0 Grade ≥ 3), any history or anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma);
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.

Sexually active males and females (of childbearing potential) unwilling to practice contraception (barriere contraceptive measure or oral contraception) during the study and until 6 months after the last trial treatment.

* Known alcohol or drug abuse;
* History of uncontrolled intercurrent illness included but not limited to:

  1. Hypertension uncontrolled by standard therapies (not stabilized to 150/90 mmHg or lower);
  2. or, uncontrolled active infection requiring antibiotics at the time of initiation of study treatment.
* Clinically significant (i.e., active) cardiovascular disease for example cerebrovascular accidents (≤6 months), transient ischemic attack, myocardial infarction (≤6 months), severe/unstable angina, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication (including correct QT interval [QTc] prolongation of > 470 msec calculated according to Fridericia and/or pacemaker or prior diagnosis of congenital long QT syndrome), or symptomatic pulmonary embolism;
* Uncontrolled coagulopathy;
* Lack of upper gastrointestinal tract integrity or malabsorption syndrome; active inflammatory bowel disease (i.e., patients requiring current medical interventions or who are symptomatic).
* All other significant disease which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment;
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent and that would limit compliance with trial requirements;
* Administration of a live, attenuated vaccine within 4 weeks prior to start of study treatment or anticipation that such a live attenuated vaccine will be required during the study. Note: administration of inactivated vaccines is allowed (for example, inactivated influenza vaccines);
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumour necrosis factor [TNF] agents) within 2 weeks prior to start of study treatment, or requirement for systemic immunosuppressive medications during the trial. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed;
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or five half-lives of the drug, whichever is longer, prior to start of study treatment;
* Legal incapacity or limited legal capacity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | 19 months
  Progression-free survival is defined as the time from enrollment to the first documentation of objective disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Toxicity Rate | 24 months
  Toxicity Rate is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing a specific adverse event of grade 3/4, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during the induction and the maintenance phases of treatment.
Objective Response Rate | 19 months
  Objective Response Rate is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria, during the induction and the maintenance phases of treatment. The determination of clinical response will be based on investigator reported measurements. Responses will be evaluated every 8 weeks.
Immuno-related Objective Response Rate | 19 months
  Immuno-related Objective Response Rate is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to immune-modified RECIST criteria, during the induction and the maintenance phases of treatment. The determination of clinical response will be based on investigator reported measurements. Responses will be evaluated every 8 weeks.
Early Objective Response Rate | up to 2 months from randomization
  Early Objective Response Rate is defined as the percentage of patients, relative to the total of the enrolled subjects, achieving a ≥ 20% decrease in the sum of diameters of RECIST target lesions at week 8 compared to baseline.
Deepness of Response | 19 months
  Deepness of Response is defined as the relative change in the sum of longest diameters of RECIST target lesions at the nadir, in the absence of new lesions or progression of non-target lesions, when compared with baseline.
R0 Resection Rate | 19 months
  R0 Resection Rate is defined as the percentage of patients, relative to the total of enrolled subjects, undergoing secondary R0 resection of metastases. Secondary R0 surgery is defined as microscopically margin free complete surgical removal of all residual disease, performed during treatment or after its completion, allowed by tumoral shrinkage and/or disappearance of one or more lesions.
Overall survival | 48 months
  Overall survival is defined as the time from registration to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Oncologia Medica 2 Universitaria - Azienda Ospedaliero-Universitaria Pisana Dipartimento di Ricerca Traslazionale e Nuove Tecnologie - University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No